CLINICAL TRIAL: NCT00568802
Title: A Pilot Therapeutic Trial Using Hydroxyurea in Type II and Type III Spinal Muscular Atrophy Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SU-11012007-781; 79233; NCT00084006 (obsolete NCT alias)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Hydroxyurea

ARMS (2):
- Hydroxyurea (Experimental)
  Interventions: Drug: Hydroxyurea
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo to match hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea
  Arms: Hydroxyurea
Drug: Placebo to match hydroxyurea
  Arms: Placebo

SUMMARY:
The objectives of this trial are: to establish a safety profile for use of Hydroxyurea in children with Types II and III Spinal Muscular Atrophy; to identify reliable outcome measures for HU treatment in Types II and III SMA; and to detect the clinical efficacy of HU treatment in children with Types II and III SMA.

DETAILED DESCRIPTION:
SMA is a neuromuscular disorder characterized by degeneration of spinal cord motor neurons and muscular atrophy. SMA is classified into three clinical subtypes according to the severity and age of onset (Types I, II and III). Type II (intermediate) SMA has its onset in early childhood (prior to 18 months) and is characterized by the failure to stand or walk unassisted. Individuals with Type III SMA (mild SMA or Kugelberg-Welander disease) typically develop symptoms after 18 months of age and display a wide range of clinical heterogeneity. The clinical spectrum ranges from rapid progressive weakness resulting in wheelchair dependence in late childhood to patients being able to walk in adult years and living productive and independent lifestyles for the majority of their lives.

In our laboratory, our preliminary results indicate that HU treatment significantly increases both SMN mRNA expression and intact SMN protein levels in vitro. These data confirm previous observations that in vitro treatments of SMA lymphocytes with hydroxyurea resulted in augmentation of the SMN2 gene expression in a dose and time related manner. Based on these exciting pre-clinical data, coupled with the well-documented side-effect profile of HU in children, we are conducting a pilot clinical trial using HU in children with Types II and III SMA. This clinical trial study is intended to establish the safety profile in children with Types II and III SMA; to identify reliable outcome measures; and to detect the possible clinical efficacy of HU treatment in children with Types II and III SMA.

ELIGIBILITY:
Inclusion Criteria:1. Laboratory confirmation of a homozygous deletion or mutation of the SMN1 gene 2. (Type II) Can sit independently but cannot walk without support by the age of 16 months and never achieve independent walking thereafter; OR (Type III) Can walk independently within the first 2 years of life, but showing rapid progression of weakness resulting in the loss of independent ambulation by 6 years of age 3. Patient is older than 16 months and younger than 8 years old at the time of enrollment

Exclusion Criteria:1. Known hematological disorders, other systemic disorders, or severe birth asphyxia 2. Participation in SMA clinical trials for other experimental drugs 3. Requiring continuous respiratory support before the initiation of HU treatment

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ching H. Wang, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data are presented for all participants because data relating to arm assignment are no longer accessible; the Principal Investigator (PI) has left institution and all efforts to locate the data have been exhausted.
Groups:
- All Participants: Participants received hydroxyurea, or placebo to match hydroxyurea.
Period: Overall Study
Arm/Group | All Participants
Started | 27
Completed | 24
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Data are presented for all participants because data relating to arm assignment are no longer accessible; the PI has left institution and all efforts to locate the data have been exhausted.
Arm/Group | All Participants
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Functional Motor Testing, Including Gross Motor Function Measure (GMFM) and Timed Motor Tests
Time Frame: Up to 6 years, 2 months
Population: Data for this outcome measure are no longer accessible; the PI has left institution and all efforts to locate the data have been exhausted.
Groups:
- Hydroxyurea: Hydroxyurea
- Placebo: Placebo to match hydroxyurea
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Safety: Frequency of Adverse Events/Lab Abnormalities
Time Frame: Up to 6 years, 2 months
Population: as for outcome 1
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pulmonary Function Testing
Time Frame: Up to 6 years, 2 months
Population: as for outcome 1
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Motor Unit Number Estimation (MUNE)
Time Frame: Up to 6 years, 2 months
Population: as for outcome 1
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Biomarker Assays: SMN Protein and SMN mRNA
Time Frame: Up to 6 years, 2 months
Population: as for outcome 1
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 years, 2 months
Description: Adverse events data are no longer accessible; the PI has left institution and all efforts to locate the data have been exhausted.
Arm/Group | Hydroxyurea | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes